CLINICAL TRIAL: NCT05443035
Title: Evaluation of Antimicrobial Photodynamic Therapy and Minimal Intervention Associated With Deproteinization in Permanent Teeth With Molar Incisor Hypomineralization: Study Protocol for a Clinical, Controlled, Blinded Trial.
Brief Title: Evaluation of Antimicrobial Photodynamic Therapy and Minimal Intervention Associated With Deproteinization in Permanent Teeth With Molar Incisor Hypomineralization
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AmandaHMI
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Hypomineralization Molar Incisor
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An independent assessor blinded to the allocation to the different groups will perform evaluations after 48 hours and at three-month intervals for a follow-up period of 12 months.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Antimicrobial PDT and Papacarie Deproteination Group (Experimental): The participants will receive selective chemical-mechanical removal of carious dentinal tissue around the walls of the cavity using a curette, followed by the application of antimicrobial PDT and deproteination with Papacárie DuoTM.
  Interventions: Procedure: Antimicrobial PDT and Papacarie Deproteinization
- Antimicrobial PDT group and deproteination with NaClO 5% group (Experimental): The participants will receive selective removal of carious dentinal tissue using a curette, followed by application of antimicrobial PDT and deproteination with NaClO 5%.
  Interventions: Procedure: Antimicrobial PDT and 5% NaOCl Deproteinization
- Control group (Experimental): The participants will receive selective removal of carious dentinal tissue using a curette.
  Interventions: Procedure: Conventional caries treatment

INTERVENTIONS:
Procedure: Antimicrobial PDT and Papacarie Deproteinization — Selective removal of carious tissue with curette + antimicrobial PDT (methylene blue 5 Evilux, Color index 52015, Fórmula & Ação + red laser at 660 nm) + deproteinization of enamel with Papacárie DuoTM + restoration.
  Arms: Antimicrobial PDT and Papacarie Deproteination Group
Procedure: Conventional caries treatment — Selective removal of carious tissue with curette + restoration.
  Arms: Control group
Procedure: Antimicrobial PDT and 5% NaOCl Deproteinization — Selective removal of carious tissue with curette + application of methylene blue and low-level laser (aPDT) + deproteinization of adjacent enamel with 5% NaOCl + restoration.
  Arms: Antimicrobial PDT group and deproteination with NaClO 5% group

SUMMARY:
Introduction: Molar Incisor Hypomineralization (MIH) is a qualitative defect of enamel development that occurs in the mineralization phase. MIH affects one or more permanent molars and, occasionally, permanent incisors. The aim of the proposed study is to evaluate the clinical effect of antimicrobial photodynamic therapy (aPDT) on permanent teeth with MIH through decontamination and sensitivity control. The longevity of the restorations will also be evaluated after the deproteinization procedure. Methods and analysis: Patients 8 to 12 years of age with permanent molars will be randomly allocated to three groups. Group 1: selective chemical-mechanical removal of carious dentinal tissue around the walls of the cavity with Papacárie Duo and a curette followed by the application of aPDT and deproteinization with Papacárie Duo; Group 2: selective removal of carious dentinal tissue around the walls of the cavity with a curette, followed by the application of aPDT and deproteinization with a 5% sodium hypochlorite solution; Group 3: selective removal of carious dentinal tissue using a curette. The selected teeth must have a carious lesion in the dentin and post-eruptive enamel breakdown on one or more surfaces with an indication for clinical restorative treatment. The teeth will subsequently be restored using a mixed technique with resin-modified glass ionomer cement and bulk-fill composite resin. The data will be submitted to descriptive statistical analysis. Associations with age and sex will be tested using either the chi-squared test or Fisher's exact test. Pearson's correlation coefficients will be calculated to determine the strength of correlations between variables. Comparisons of the microbiological results (colony-forming units) will be performed using ANOVA and the Kruskal-Wallis test. Kaplan-Meier survival analysis will be performed to assess the performance of the restorations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children with no adverse systemic conditions;
* At least one permanent first molar with MIH and active caries on the dentin with post-eruptive fracture on a single surface or multiple surfaces with an indication for restorative treatment; direct view and access; no clinical or radiographic signs or symptoms of pulpal involvement;
* Hypomineralized enamel with opacities near the margins of the cavities;
* Occurrence or non-occurrence of dentinal sensitivity.

Exclusion Criteria:

* Clinically: carious lesion only involving the enamel, deficient restorations, small carious lesions in dentin (without access to manual excavator), hidden caries, clinical sign or symptom of pulpal involvement, clinical impossibility of restoration;
* Radiographically: evidence of pulpal involvement;
* Teeth severely affected by MIH without indication for restorative treatment;
* Partially erupted teeth with MIH.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 69 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-03-20 (Estimated)

PRIMARY OUTCOMES:
Change in retention of the restorative material in the cavity | 48 hours after the restorative treatment and at three-months intervals for a period of 12 months of follow up.
  The effects of deproteination on the longevity of the restoration will be evaluated using the modified USPHS index, in which retention, marginal integrity, marginaldiscoloration, anatomic form and secondary caries are evaluated.

SECONDARY OUTCOMES:
Change in microbiological evaluation | Baseline and immediately after treatment.
  Prior to the removal of the carious tissue, a sample infected dentin will be collected from each selected tooth. Immediately after the removal of the carious tissue and the application of aPDT, a sample of the remaining dentin will be collected. The results will be expressed as colony-forming units of SM and LB as well as proportion of streptococci (% S/TM), streptococci of the mutans group (% SM/TM) and lactobacilli (% LB/TM) in relation to the total of viable microorganisms. For SM, the proportion in relation to the total of streptococci (% SM/S) will also be calculated.
Change in Dental Sensitivity | Baseline, 48 hours after the restorative treatment and at three-months intervals for a period of 12 months of follow up.
  Prior to the removal of the carious tissue, the volunteers in the different groups will indicate the degree of pain or discomfort on the visual analog scale (VAS) following isolation of the neighboring teeth and the application of compressed air to the tooth with MIH for 3 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Nove de Julho University, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The information collected from the participants will be transcribed into a database replacing the individuals' names with the registration number of the evaluation form. The datasets (Excel spreadsheets) generated from this protocol will be available from the corresponding author (Sandra Kalil Bussadori - sandra.skb@gmail.com) upon any reasonable request. However, reuse of this data will not be permitted for anyone who is not an author of this paper.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available as soon as the article with the findings will be published in a peer-reviewed journal.
Access Criteria: The datasets from this protocol will be available from the corresponding author (Sandra Kalil Bussadori -sandra.skb@gmail.com) upon any reasonable request.

REFERENCES:
- [Derived] Mandetta ARH, Bortoletto CC, Sobral APT, Goncalves MLL, Motta LJ, Horliana ACRT, Ferrari RAM, Prates RA, Deana AM, Cordeiro RCL, Pinto LAMDS, Fernandes KPS, Bussadori SK. Evaluation of antimicrobial photodynamic therapy and minimal intervention associated with deproteinisation in permanent teeth with molar incisor hypomineralisation: study protocol for a clinical, controlled, blinded trial. BMJ Open. 2023 Dec 14;13(12):e076226. doi: 10.1136/bmjopen-2023-076226. PMID 38101830